CLINICAL TRIAL: NCT00314054
Title: An Open-Label, Single-Dose, Parallel-Group Study of the Pharmacokinetics and Safety of HCV-796 in Subjects With Chronic Hepatic Impairment and in Matched Healthy Adults
Brief Title: Study Evaluating the Safety of HCV-796 in Subjects With Liver Disease and in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Collaborators: ViroPharma (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3173A1-105
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Last update posted 2008-04-14 (Estimated); Status verified 2008-04

CONDITIONS: Hepatitis C; Hepatic Insufficiency
Keywords: Hepatitis C; Hepatic Impairment; Healthy Volunteer; Phase 1; Hepacivirus
MeSH Terms: conditions — Hepatitis C; Hepatic Insufficiency | interventions — HCV 796

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): HCV-796 1000mg single dose
  Interventions: Drug: HCV-796

INTERVENTIONS:
Drug: HCV-796 — HCV-796 1000mg single dose

SUMMARY:
The purpose of this study is to assess the pharmacokinetics (PK) of HCV-796 in subjects with chronic hepatic impairment and in matched healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of non-childbearing potential.
* Hepatic impairment subjects: Child-Pugh class A, B, or C according to the C-P classification based on history, physical examination, and laboratory test results.
* Healthy volunteers: healthy as determined by the investigator.

Exclusion Criteria:

* History of alcoholism within 1 year.
* Hepatic impairment subjects: evidence of unstable clinically significant disease other than impaired hepatic function.
* Healthy volunteers: positive serologic findings for hepatitis B surface antigen (HBsAg) and/or hepatitis C virus (HCV) antibodies.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2006-05; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
To assess PK in subjects with chronic hepatic impairment and in matched healthy adults | 7 days

SECONDARY OUTCOMES:
To assess the safety and tolerability in subjects with chronic hepatic impairment and in matched healthy adults | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (3):
- United States (3):
  - Gainesville, Florida
  - Orlando, Florida
  - Saint Paul, Minnesota